CLINICAL TRIAL: NCT02284958
Title: A Single-centre, Randomized Controlled Trial Investigating Clinical Utility and Cost-effectiveness of an Individualized Pedometer Driven Walking Programme for People With Chronic Low Back Pain
Brief Title: Walking Away From Back Pain, One Step at a Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: University of Ulster (Other); University of Nottingham (Other); University of Otago (Other)
Responsible Party: Principal Investigator, Stephan Milosavljevic, Principal Investigator, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-218
Record Dates: First submitted 2014-10-23; First posted 2014-11-06 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Low Back Pain
Keywords: walking; pedometer
MeSH Terms: conditions — Low Back Pain | interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard/Control group (Active Comparator): Each participant will receive a one-off individualized educational session regarding the management of chronic low back pain with a Physical Therapist: includes a physical examination, standardized advice & provision of the 'Back Book'.
  Interventions: Behavioral: Standard
- Walking group (Experimental): Each participant will receive a one-off educational session as per standard/control group followed by a 12 week graded, individually tailored, pedometer driven walking programme given by a Physical Therapist. Participants will be monitored each week and provided with encouragement and advice to increase the number of steps taken each day.
  Interventions: Behavioral: Walking

INTERVENTIONS:
Behavioral: Standard — Back care advice
  Arms: Standard/Control group
Behavioral: Walking — Back care advice, individualized 12 week pedometer-driven walking program
  Arms: Walking group

SUMMARY:
This study will investigate if a 12-week, individually-tailored walking program, using pedometers will be a more clinically and cost-effective option for the management of chronic low back pain than standardized advice and education.

DETAILED DESCRIPTION:
Specific objectives of the study are:

1. To determine perceived levels of disability and baseline levels of walking activity in a sample of those with chronic low back pain (CLBP)
2. To determine the uptake and adherence to a pedometer-driven walking program for people with CLBP
3. To test the clinical and cost-effectiveness of a walking programme to improve outcomes for CLBP compared to a standardized back care education package
4. To test the feasibility of a walking programme in a sub-sample of rural Saskatchewan farmers/agricultural workers.

ELIGIBILITY:
Inclusion Criteria:

* males and females aged 18 years or over,
* experiencing low back pain (i.e. between the 12th costal margin and gluteal fold with or without associated leg pain) persisting for a minimum of three months, and
* assessed as capable of participating in a walking programme.

Exclusion Criteria:

* any spinal surgery in the past 12 months;
* evidence of nerve root, spinal cord, or cauda equina compression;
* severe spinal stenosis indicated by signs of neurogenic claudication, grade 3 to 4 spondylolisthesis, fibromyalgia, or systemic/inflammatory disorder;
* as well as any other current lower extremity musculoskeletal injury or contraindication to increasing physical activity (PA) levels.

The latter may include:

* any cardiorespiratory or other medical condition limiting exercise tolerance;
* history of serious psychological or psychiatric illness (mild depression eligible for inclusion); and/or
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2015-04; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in Oswestry Low Back Pain Disability Questionnaire score | Baseline, 12 weeks, 6 months and 12 months

SECONDARY OUTCOMES:
Change in mean number of steps per day for each week of the study | Baseline & 12 weeks
Change in six minute walk test | Baseline, 12 weeks, 6 months & 12 months
Change in International Physical Activity Questionnaire score | Baseline, 12 weeks, 6 months & 12 months
Change in Fear Avoidance Beliefs Questionnaire score | Baseline, 12 weeks, 6 months & 12 months
Change in Back Beliefs Questionnaire score | Baseline, 12 weeks, 6 months & 12 months
Change in Exercise Self-efficacy Scale score | Baseline, 12 weeks, 6 months & 12 months
Change in Global rating of change for physical activity score | Baseline, 12 weeks, 6 months & 12 months
Change in Euroqual-5D score | Baseline, 12 weeks, 6 months & 12 months
  Quality of life
Change in health care usage and intervention costs over time | Baseline, 12 weeks, 6 months & 12 months
  Participant records health care usage and intervention costs over the 12 month study
Focus group data | Following 12 week intervention
  Walking group only, voluntary participation

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Milosavljevic, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Derived] Lang AE, Hendrick PA, Clay L, Mondal P, Trask CM, Bath B, Penz ED, Stewart SA, Baxter GD, Hurley DA, McDonough SM, Milosavljevic S. A randomized controlled trial investigating effects of an individualized pedometer driven walking program on chronic low back pain. BMC Musculoskelet Disord. 2021 Feb 19;22(1):206. doi: 10.1186/s12891-021-04060-8. PMID 33607979
- [Derived] Milosavljevic S, Clay L, Bath B, Trask C, Penz E, Stewart S, Hendrick P, Baxter GD, Hurley DA, McDonough SM. Walking away from back pain: one step at a time - a community-based randomised controlled trial. BMC Public Health. 2015 Feb 13;15:144. doi: 10.1186/s12889-015-1496-9. PMID 25885913